CLINICAL TRIAL: NCT00466089
Title: Phase II Randomized Trial of 3D Radiotherapy Versus the Combination of 3D Radiotherapy and Erlotinib (Tarceva®) in Patients With Localized-Unresectable Non-Small Cell Lung Cancer Non Susceptible for Chemotherapy Treatment.
Brief Title: Study of 3D Radiotherapy With or Without Erlotinib (Tarceva®) in Patients With Localized Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital of Navarra (Other)
Collaborators: Dr. Enrique Martínez López (Unknown)
Responsible Party: Dr. Enrique Martínez López, Dr. Enrique Martínez López
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO19182
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC, lung cancer; Patients with localized-unresectable (IA-IIIB) non-small cell lung cancer non susceptible for chemotherapy treatment.
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): RT + Tarceva
  Interventions: Drug: Erlotinib (Tarceva®)
- 2 (No Intervention): RT

INTERVENTIONS:
Drug: Erlotinib (Tarceva®) — Erlotinib (Tarceva®), 150mg/day p.o during 6 months.
  Arms: 1

SUMMARY:
A phase II, multicenter, randomized trial of 3D Radiotherapy versus 3D Radiotherapy and erlotinib (Tarceva®) in patients with localized-unresectable (IA-IIIB) non-small cell lung cancer non susceptible for chemotherapy treatment, to compare safety and toxicity profile, and the progression-free survival in both arms of treatment (3D Radiotherapy versus 3D Radiotherapy + erlotinib) in patients who have not received previous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any specific procedure of the protocol.
* Histologically confirmed diagnosis of non small cell lung cancer.
* Unresectable (IA-IIIB) non-small cell lung cancer.
* Patients non susceptible for chemotherapy treatment
* Measurable disease according to RECIST criteria
* Age > 18 years.
* ECOG performance status < 2.
* Adequate bone marrow, hepatic, renal and respiratory function.
* Patients capable of following an adequate therapeutic compliance and accessible for a correct follow-up.
* Women at a fertile age must have a negative serum or urine pregnancy test within the 7 days prior to the beginning of the treatment.
* Patients of both genders at a fertile age, including those women having their last menstruation within the two previous years, must follow effective contraceptive measures.

Exclusion Criteria:

* Prior chemotherapy or radiotherapy.
* History of other curatively treated malignancy and no evidence of disease within the past 5 years except squamous cell skin cancer, or resected cervix carcinoma.
* Pregnant or lactating women.
* Any other severe disease or clinical conditions, as, but not only:

  1. Unstable cardiopathy despite treatment, myocardial infarction within the 6 months before entering the study
  2. Uncontrolled active infection
  3. Uncontrolled peptic ulcer, unstable diabetes mellitus or any other contraindication for treatment with corticosteroids.
  4. Autoimmune diseases.
* Concomitant treatment with any other antineoplastic therapy.
* Prior experimental pharmacological agent within the 3 weeks prior to the inclusion of the study.
* Prior treatment with EGFR targeted therapies.
* Erlotinib known hypersensibility.
* Any radiotherapy treatment contraindication.
* History of significant neurological or psychiatric disorders, including epileptic seizures.
* Any significant ophthalmologic impairment of the eye surface (Use of contact lenses is not recommended)
* Inability to take oral medication and surgical procedures affecting the absorption or implying intravenous or parenteral feeding.
* Any other underlying severe process affecting the ability to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-03

PRIMARY OUTCOMES:
To determinate the viability and toxicity profile of Erlotinib + 3D Radiotherapy treatment (% of patients presenting toxicity 3-4 during the treatment).

SECONDARY OUTCOMES:
The progression-free survival.
1-year survival.
Overall survival.
Objective response rate, according to RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Martínez, Dr., Principal Investigator — Hospital de Navarra; Ana Mª Perez Casas, Dr., Principal Investigator — Fundación Jimenez Diaz; Alejandro De la Torre, Dr., Principal Investigator — Hospital Puerta de Hierro; Francesc Casas, Dr., Principal Investigator — Hospital Clínic i Provincial de Barcelona; Nuria Viñolas, Dr., Principal Investigator — Hospital Clínic i Provincial de Barcelona; Julian Minguez, Dr., Principal Investigator — Hospital de Donostia
Locations (5):
- Spain (5):
  - Hospital Clínic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Fundación Jimenez Diaz, Madrid, Madrid
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital de Donostia, Donostia / San Sebastian, San Sebastian